CLINICAL TRIAL: NCT06977529
Title: The Effect Of Algorithm-Guided Care Provided To Total Knee Prosthesis Patients On Fall And Recovery: Randomized Controlled Trial
Brief Title: Fall Prevention in Total Knee Replacement Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Sibel ARSLAN, Assistant Professor, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Gaziantep Unıv.
Record Dates: First submitted 2025-03-24; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Total Knee Arthroplasty
Keywords: ALGORİTHM; FALL; PATİENT SAFETY; TOTAL KNEE ARTHROPLASTY
MeSH Terms: interventions — Algorithms; Early Ambulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERİMENTAL (Experimental): The "Fall Prevention Algorithm" prepared by the researchers was applied to the experimental group patients.
  Interventions: Behavioral: Algorithm; Algorithm-based maintenance created by researchers:such as falls training, early mobilization
- control (No Intervention): No intervention was made by the researcher.

INTERVENTIONS:
Behavioral: Algorithm; Algorithm-based maintenance created by researchers:such as falls training, early mobilization — The "Fall Prevention Algorithm" prepared by the researchers was applied to the experimental group patients.
  Arms: EXPERİMENTAL

SUMMARY:
Falls, one of the patient safety goals, lead to injury and death if not prevented. This study was conducted to determine the effect of algorithm-guided care on falling, fear of movement, fear of falling and postoperative recovery index for patients with total knee replacement surgery at high risk of falling. The research was conducted as a randomized, controlled and experimental study in the orthopedic clinics of a city hospital and a state hospital between 20.01.2024 and 04.06.2024. The sample of the study consisted of 56 patients who would undergo total knee replacement surgery with a high risk of falling. The patients were divided into two groups: experimental (n=28) and control (n=28) groups. "Patient Questionnaire", "Postoperative Recovery Index (ASII)", "Tampa Kinesiophobia Scale (TKÖ)", "International Fall Effectiveness Scale (UDES)" were applied to all patients participating in the study. The "Fall Prevention Algorithm" prepared by the researchers was applied to the experimental group patients.

ELIGIBILITY:
Inclusion Criteria:

* Having a unilateral total knee replacement surgery for the first time,
* Not having a psychiatric illness diagnosis,
* Being able to speak and understand Turkish,
* Being willing to participate in the research.

Exclusion Criteria:

* Patients who will undergo emergency surgery,
* Have hearing and speech problems,
* Have visual impairment,
* Have conditions that may affect cognitive functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
FALL | Perioperative period , Within 30 days after surgery.
  Patients' fall status will be recorded by asking questions in the "Patient Questionnaire Form".

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Universty, Gaziantep, ŞAHİNBEY, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No